CLINICAL TRIAL: NCT01689714
Title: A MULTI-CENTER CLINICAL STUDY TO EVALUATE THE SAFETY AND EFFICACY OF FOLATESCAN (TECHNETIUM Tc 99m EC20) IN PATIENTS WITH SUSPECTED OVARIAN CARCINOMA OR RECURRENT ENDOMETRIAL CARCINOMA
Brief Title: Safety and Efficacy of Folatescan (Technetium TC 99M EC20) in Patients With Suspected Ovarian Carcinoma or Recurrent Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.4
Record Dates: First submitted 2012-09-09; First posted 2012-09-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-09

CONDITIONS: Ovarian Carcinoma; Recurrent Endometrial Carcinoma
Keywords: Ovarian Carcinoma; Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tc 99m EC20 (Experimental): Patients received 2 intravenous (IV) injections: 1 mg of folic acid (to reduce the uptake of FolateScan in normal tissues), followed 1 to 3 minutes later by 0.1 mg of EC20 labeled with 15 to 25 mCi of technetium-99m (99mTc) over 30 seconds in a total injection volume of 1 to 2 mL.2 Each injection was given as a slow IV push via a free-flowing indwelling IV catheter in an upper extremity vein (i.e., in the antecubital fossa).
  Interventions: Drug: Tc 99m EC20

INTERVENTIONS:
Drug: Tc 99m EC20

SUMMARY:
The folate receptor is overexpressed in many types of cancer, including ovarian and endometrial cancer, and the level of folate receptor expression increases with the stage of the disease. Technetium Tc 99m EC20 (99mTc-EC20; FolateScan), a folate-targeted diagnostic radiopharmaceutical, is designed to bind to the folate receptor. Thus, FolateScan may provide an effective method to determine folate receptor-positive (FR+) target tumors, thereby assisting in the identification of those patients who may benefit from folate-targeted therapy.

DETAILED DESCRIPTION:
This phase 2, two-center, open-label, single-treatment group, within-patient-controlled study was conducted to:

* Expand the safety database and gather data on the percentage of patients with known or suspected ovarian carcinoma or recurrent endometrial carcinoma who show increased uptake of FolateScan in tumors (primary objective).
* Calculate the sensitivity, specificity, accuracy, positive predictive value, and negative predictive value of FolateScan compared with immunohistochemical (IHC) staining (secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following eligibility requirements to be enrolled in the study.

  1. Subject must be 18 years of age or older.
  2. Subject must have known or strongly suspected ovarian carcinoma or recurrent endometrial carcinoma with at least one identifiable lesion > 1.5 cm as diagnosed by ultrasonography, MRI, or CT.
  3. Subject must have good kidney function.
  4. Subject must provide written informed consent prior to enrollment.

Exclusion Criteria:

* Subjects must be excluded if any of the following conditions are present:

  1. Subject is pregnant or breastfeeding.
  2. Subject is simultaneously participating in another investigational drug study.
  3. Subject has completed the follow-up phase of any previous study less than 30 days prior to enrollment in this study.
  4. Subject is unable to tolerate conditions for radionuclide imaging.
  5. Subject has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-08; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Val J Lowe, MD, Principal Investigator — Mayo Clinic